CLINICAL TRIAL: NCT02596555
Title: Safety and Efficacy of Low Molecular Weight Heparin for 72 Hours Followed by Dabigatran for the Treatment of Acute Intermediate-Risk Pulmonary Embolism
Brief Title: Low Molecular Weight Heparin for 72 Hours Followed by Dabigatran for Acute Intermediate-Risk Pulmonary Embolism.
Acronym: PEITHO-2
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: 1. Interim results suggested a reduction of sample size.
  2. Anticipated length of enrolment period with resulting funding issues to pose a threat to the study.
Sponsor: Prof. Stavros Konstantinides, MD (Other)
Collaborators: European Georges Pompidou Hospital (Other)
Responsible Party: Sponsor-Investigator, Prof. Stavros Konstantinides, MD, Medical Director of Center for Thrombosis and Hemostasis, University Medical Center Mainz, Johannes Gutenberg University Mainz
Organization: Johannes Gutenberg University Mainz (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEITHO-2
Record Dates: First submitted 2015-11-03; First posted 2015-11-04 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — Dabigatran

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dabigatran treatment (Experimental): Low molecular weight heparin for 72 hours followed by 6 months of dabigatran
  Interventions: Drug: Dabigatran

INTERVENTIONS:
Drug: Dabigatran — Low molecular weight heparin for 72 hours followed by 6 months of dabigatran
  Other Names: Pradaxa

SUMMARY:
This prospective, multicenter, multinational, phase IV, interventional single-armed (management) trial will focus on the safety, efficacy and cost-effectiveness of a new oral anticoagulant in the treatment of patients with acute intermediate-risk PE based on validated imaging (echocardiographic or CT angiographic) and laboratory biomarker (circulating levels of cardiac troponins and natriuretic peptides) parameters and their combinations.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Objectively confirmed diagnosis of acute PE by multidetector CT angiography, ventilation/perfusion lung scan, or selective invasive pulmonary angiography, according to established diagnostic criteria, with or without symptomatic deep vein thrombosis
3. Absence of hemodynamic collapse, or decompensation, at presentation; Hemodynamic collapse or decompensation
4. Intermediate-risk category of PE severity indicated by a positive (score ≥1) simplified pulmonary embolism severity index (sPESI), in combination with the presence of at least one of the following criteria at presentation:

   * At least one sign of RV pressure overload/dysfunction on CT angiography or echocardiography
   * Signs of myocardial injury as indicated by elevated troponin levels
   * Signs of (RV) failure as indicated by NT-proBNP levels >600 pg/ml at baseline.
5. Ability of the subject to understand the character and individual consequences of the clinical trial; signed and dated informed consent of the subject available before the start of any specific trial procedures

Exclusion Criteria:

1. Pregnancy (a negative serum or urine pregnancy test should be available for women of child-bearing potential before study inclusion) or lactation
2. Women of childbearing potential who do not practice a medically accepted highly effective contraception during the trial and one month beyond
3. History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product
4. Participation in another clinical trial during the present clinical trial or within the last three months
5. Medical or psychological condition that would not permit completion of the trial or signing of informed consent
6. Use of a fibrinolytic agent, surgical thrombectomy, interventional (catheter-directed) thrombus aspiration or lysis, or use of a cava filter to treat the index episode of PE
7. Treatment with any therapeutically dosed anticoagulant for more than 48 hours prior to enrolment
8. Need for long-term treatment with a low molecular weight heparin, vitamin K antagonists or NOAC, for an indication other than the index PE episode, or for antiplatelet agents except acetylsalicylic acid at a dosage ≤100 mg/day;
9. Active bleeding or known significant bleeding risk (e.g., gastrointestinal ulcer, malignant neoplasms, injuries or recent surgeries of the brain, spinal cord or eyes, recent intracranial bleedings, known or suspected esophagus varices, aneurysms or intraspinal or intracranial vascular abnormalities)
10. Artificial heart valves requiring treatment with an anticoagulant
11. Renal insufficiency with estimated creatinine clearance <30 ml/min/1.73m2
12. Chronic liver disease with aminotransferase levels two times or more above the local upper limit of normal range
13. Concomitant administration of strong inhibitors of P-glycoprotein like ketoconazole, cyclosporin, itraconazole or dronedarone
14. Unwillingness or inability to adhere to treatment or to the follow-up visits
15. Life expectancy less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Occurrence of symptomatic venous thromboembolism (VTE) or pulmonary embolism (PE) related death (yes/no) | 6 months

SECONDARY OUTCOMES:
Recovery of right ventricle (RV) function | 6±1 days or upon discharge (whichever comes first), 6 months
Temporal pattern of changes in NT-proBNP (N-terminal prohormone of brain natriuretic peptide) levels | 6±1 days or upon discharge (whichever comes first), 6 months
Death from any cause | 30 days
Pulmonary embolism (PE) related death, or PE-related or hemodynamic collapse or decompensation | 30 days
Overall duration of hospital stay | 6 months
Major bleeding | 6 months
Clinically relevant bleeding | 6 months
Serious adverse events (SAE) | 72 hours, 30 days, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Konstantinides, Prof., MD, Principal Investigator — Center for Thrombosis and Hemostasis, University Medical Center Mainz
Locations (1):
- Center for Thrombosis and Hemostasis, University Medical Center Mainz, Mainz, Germany

REFERENCES:
- [Derived] Klok FA, Toenges G, Mavromanoli AC, Barco S, Ageno W, Bouvaist H, Brodmann M, Cuccia C, Couturaud F, Dellas C, Dimopoulos K, Duerschmied D, Empen K, Faggiano P, Ferrari E, Galie N, Galvani M, Ghuysen A, Giannakoulas G, Huisman MV, Jimenez D, Kozak M, Lang IM, Lankeit M, Meneveau N, Munzel T, Palazzini M, Petris AO, Piovaccari G, Salvi A, Schellong S, Schmidt KH, Verschuren F, Schmidtmann I, Meyer G, Konstantinides SV; PEITHO-2 investigators. Early switch to oral anticoagulation in patients with acute intermediate-risk pulmonary embolism (PEITHO-2): a multinational, multicentre, single-arm, phase 4 trial. Lancet Haematol. 2021 Sep;8(9):e627-e636. doi: 10.1016/S2352-3026(21)00203-9. Epub 2021 Aug 4. PMID 34363769